CLINICAL TRIAL: NCT06559579
Title: Comparative Study of Clinical Disorders Related to Monoclonal Gammopathy in Patients With Haematological Malignancies in Two Hospitals in Finistère Between 2012 and 2017 (GammaClinik)
Brief Title: Monoclonal Gammopathy With Clinical Significance in Patients With and Without Haematological Malignancies in Finistère Between 2012 and 2017 (GammaClinik)
Acronym: GammaClinik
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0282 - GammaClinik
Record Dates: First submitted 2023-08-03; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Gammopathy, Monoclonal
MeSH Terms: conditions — Paraproteinemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical symptoms associated with monoclonal gammapathy have been primarily studied in hematological malignancy and rarely in MGUS and hemopathy. Indeed, most studies focus on a specific type of clinical involvement that does not allow to understand the epidemiological distribution of clinical symptoms in this population. In addition, in most cases, studies of clinical impairment of monoclonal gammapathies focus on one symptom. This study could highlight disparities in the representation of clinical disorders associated with monoclonal gammapathies, depending on whether they are or not associated with a malignant hematology, and would provide a better overall picture of the distribution of these diseases. This study could potentially define prognosis values for certain clinical conditions that we would not find in the group of hematological malignancies. This study would also make it possible to investigate whether there are clinical disorders of monoclonal gammapathies associated with chronic lymphoma/lymphocytic leukemia. This would potentially guide future pathophysiological research. This bicentric study could, depending on the results, be supplemented later by a larger study.

ELIGIBILITY:
Inclusion Criteria:

ge > 18 years Patient with monoclonal gammapathy of undetermined significance with clinical involvement associated with gammapathy or a malignant hematology (myeloma, plasmocytoma, Waldenström's disease, chronic lymphocytic leukemia, B lymphoma) with a monoclonal peak responsible for clinical impairment, Diagnosis of either monoclonal peak, haematopathy or clinical involvement between 2012 and 2017 Obtaining the non opposition

NB: Clinical Impairment:

* Amylose AL
* cryoglobulinemia
* acquired inhibitor C1 deficiency
* Acquired Willebrand disease;
* bullous dermatosis
* xanthomatosis and xanthogranulomatosis neccrobiotic
* Cold agglutinin disease;
* peripheral neuropathy (anti MAG neuropathy, anti ganglioside, CANOMAD)
* hemolytic uremic syndrome and PTT
* anomaly alternate route of complement
* POEMS syndrome
* Capillary leak and clarkson syndrome
* TEMPI syndrome
* neutrophilic dermatosis: sweet syndrome, sneddon and wilkinson corneal pustulosis, erythema elvatum diutinum, pyoderma gangrenosum
* cutis laxa acquis
* mucinopapulosis
* Schnitzler
* myopathy (Sporadic Late Onset Nemaline Myopathy)
* idiopathic thrombocytopenic purpura
* autoimmune hemolytic anemia
* hyperparathyroidia
* amyotrophic lateral sclerosis
* myasthenia
* Overload crystalline histiocytosis
* Crystalline keratopathy
* GOMMID (monoclonal immunoglobulin microtubular organized deposition glomerulonephritis)
* immunotactoid glomerulopathy
* fanconi syndrome
* randall disease
* PGNMID (Monoclonal immunoglobulin light-chain non-Organic glomerulonephritis)
* Glomerular basal anti-membrane disease
* Extramembranous glomerulonephritis
* glomerulonephritis with C3 deposition

Exclusion Criteria:

* Clinical involvement due to another condition of the patient (diabetes, hypertension, etc.) Clinical involvement due to chemotherapy Clinical involvement due to a strong tumor mass (IgM cutaneous deposition in Waldenström, cylindrical myeloma nephropathy, hyperviscosity syndrome in Waldenström) Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with monoclonal gammopathy of indeterminate significance (MGUS) or malignant hematology (myeloma, plasmocytoma, Waldenström disease, chronic lymphoid leukemia, B lymphoma), diagnosed between 2012 and 2017 and associated with a monoclonal gammopathy and clinical impairment within the spectrum of clinically significant gammopathy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Search for a difference in the distribution of the various clinical conditions associated with monoclonal peaks in gammapathies of undetermined significance compared with hematological malignancies. | 5 years
  The presence of a difference in the distribution of gammopathy-related clinical disorders between GMSI and hemopathies

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Brest, Brest
  - CHIC de Quimper, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.